CLINICAL TRIAL: NCT07290374
Title: Mckenzie Versus Maitland Cervical Mobilization Technique in Management of Non-specific Neck Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Salah Abd-Elfattah, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/006047
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: Maitland; Mckenzie; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mckenzie exercises group (Experimental): This group will receive Mckenzie exercises and the conventional treatment 3 sessions per week for four weeks
  Interventions: Other: Mckenzie exercises
- Maitland mobilization for cervical spine group (Experimental): This group will receive Maitland mobilization for cervical spine and the conventional treatment 3 sessions per week for four weeks
  Interventions: Other: Maitland mobilization for cervical spine
- The onventional treatment group (Active Comparator): This group will receive only the conventional treatment 3 sessions per week for four weeks
  Interventions: Other: The conventional treatment group

INTERVENTIONS:
Other: Mckenzie exercises — Fifteen participants will receive Mckenzie exercises prescribed by McKenzie for cervical dysfunction from sitting position with the following progressions:
  1. Repeated movements in the direction of the dysfunction.
  2. Repeated movements with patient overpressure.
  3. Repeated movements with therapist overpressure. All exercises will be performed while maintaining retraction position with repetition of 10 to 15 times.
  This group will also receive the conventional treatment prescribed for chronic Non-specific neck pain in the form of hot packs, postural correction, stretching, Isometric strengthening and scapular stabilization exercises.
  Arms: Mckenzie exercises group
Other: Maitland mobilization for cervical spine — Fifteen participants will receive Mailand mobilization for cervical spine: With one or two oscillations per second for one-minute, central postero-anterior (P/A) glide over spinous process in case of central or bilateral symptoms and unilateral postero-anterior (P/A) glide over articular process in case of unilateral symptoms. Grade 1 or 2 will be applied to relieve pain while grade 3 or 4 will be applied to increase ROM.
  This group will also receive the conventional treatment prescribed for chronic Non-specific neck pain in the form of hot packs, postural correction, stretching, Isometric strengthening and scapular stabilization exercises.
  Arms: Maitland mobilization for cervical spine group
Other: The conventional treatment group — Fifteen participants will receive only the conventional physical therapy program prescribed for chronic non-specific neck pain in the form of:
  1. Source of superficial heat using hot packs for 15 minutes.
  2. Postural correction exercises.
  3. Isometric strengthening exercises for neck muscles in all directions (Flexion, extension, side bending and rotation).
  4. Stretching for common tight muscles (Trapezius, levator scapulae and sternocleidomastoid muscles).
  5. Chin tuck exercises.
  6. Scapular stabilization exercises.
  Arms: The onventional treatment group

SUMMARY:
This study will be conducted to compare between Mckenzie exercises and Maitland cervical mobilization technique in management of non-specific neck pain as regard to neck pain, cervical range of motion, neck function and cervical proprioception.

DETAILED DESCRIPTION:
Neck pain is the second leading cause of disability worldwide among people with musculoskeletal disorders , and neck pain is responsible for a substantial burden to society .

Current guidelines advocate a multimodal approach including different types of exercise and manual therapy for managing non-specific neck pain and there is little evidence of what specific intervention of this multimodal approach is most beneficial. This means that there is a gap in literature regarding this point in general. If effectiveness of each intervention is clear, this will inform selection of individual components of the multimodal approach.

45 Subjects of both genders with a primary complaint of neck pain more than 12 weeks will participate in this study.Group A will receive Mckenzie exercise in the form of repeated movements in the direction of painful & restricted movement .Group B: will receive Maitland's cervical mobilization in the form of posterior-anterior (PA) glide.Group C: will receive only the conventional physical therapy program prescribed in the form of ( hot packs , stretching exercises, isometric strengthening exercises and postural correction exercises).

ELIGIBILITY:
Inclusion criteria:

* 45 Subjects diagnosed and referred from orthopedist with chronic NSNP.
* All participants will have neck pain with mobility deficit according to ICF classification of neck pain..
* Duration of symptoms is more than 3 months to be chronic.
* Subjects of both genders will be involved in the study.
* Subject are young adult with the age span between 18 &29 years because this period is characterized by extensive changes, handling choices and opportunities such as moving out from home, choice of education and career, and establishing an adult lifestyle.
* All participants will be selected with body mass index (BMI) between 18.5 and 24.9kg/cm2 which is considered the normal range of BMI.

Exclusion criteria:

* History of cervical surgery.
* Whiplash injuries.
* Inflammatory arthropathy.
* Myelopathy.
* If neck pain is associated with radiculopathy.
* Vertebrobasilar insufficiency.
* Red flags suggesting of cancer or infection .
* Fracture.
* Diabetic patients.
* Hypertensive patients.
* Obese subjects.
* Vertigo.
* Thoracic outlet syndrome.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Cervical proprioception | 4 weeks
  Cervical proprioception will be assessed using CROM device.
Cervical range of motion | 4 weeks
  Cervical ROM will be assessed using CROM device.

SECONDARY OUTCOMES:
Neck function | 4 weeks
  Arabic version of neck disability index will be used to assess neck function
Pain intensity | 4 weeks
  Numerical Rating Scale will be used to assess pain intensity

IPD SHARING:
Plan to Share IPD: No